CLINICAL TRIAL: NCT07316088
Title: Determining the Potential for Efficacy of OTX-601 in Reducing PTSD Symptoms in a Randomized Controlled Trial (RCT)
Brief Title: Determining the Potential for Efficacy of OTX-601 in Reducing PTSD Symptoms
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oui Therapeutics, Inc. (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Florida State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-Oui-002-Study2; R44MH136888 (NIH)
Record Dates: First submitted 2025-12-30; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: PTSD; Post Traumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OTX-601 (Experimental): A prescription digital therapeutic designed to overcome existing barriers and deliver evidence based treatment for PTSD
  Interventions: Device: OTX-601 Digital Therapeutic
- OTX-003 (Sham Comparator): OTX-003 is a smartphone application developed as a comparator to OTX-601 and designed to match its interface while providing no active PTSD treatment.
  Interventions: Device: OTX-003 Comparator app

INTERVENTIONS:
Device: OTX-601 Digital Therapeutic — Prescription digital therapeutic designed to overcome existing barriers and deliver evidence-based treatment for PTSD
  Arms: OTX-601
Device: OTX-003 Comparator app — Comparator designed to match interface of intervention while providing no active treatment.
  Arms: OTX-003

SUMMARY:
This study is exploring the efficacy of a digital therapeutic app in reducing symptoms of posttraumatic stress disorder (PTSD) in adults.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a randomized controlled trial to evaluate the efficacy of OTX-601 (intervention) compared to OTX-003 (comparator) in reducing PTSD symptoms from baseline to 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Posttraumatic stress disorder (PTSD) diagnosis
* Anxiety Sensitivity Index 3 (ASI-3) scores above 24
* PTSD Checklist for DSM-V (PCL-5) scores above 30
* Understands and speaks English
* Access to a smartphone that is connected to the internet

Exclusion Criteria:

* Score of 24 or lower on the ASI-3
* Score of 30 and below on the PCL-5
* No PTSD diagnosis
* Active psychosis
* Acute intoxication during study baseline
* Enrolled in another treatment research study
* Medical illness that would prevent the completion of interoceptive exposure exercises

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD symptoms between baseline and week 7 | Baseline, Week 7
  Change in PTSD symptoms will be ascertained with the PTSD Checklist for DSM-V (PCL-5). The PCL-5 total score ranges from 0 to 80, with higher scores indicating more severe symptoms.

SECONDARY OUTCOMES:
Change in PTSD symptoms at weeks 15 and 27 | Week 15, Week 27
  Change in PTSD symptoms will be ascertained with the PTSD Checklist for DSM-V (PCL-5). The PCL-5 total score ranges from 0 to 80, with higher scores indicating more severe symptoms.
Change in Anxiety Sensitivity at weeks 7, 15, and 27 | Week 7, Week 15, Week 27
  Change in Anxiety Sensitivity will be measured using the Anxiety Sensitivity Index-3 (ASI-3). The ASI-3 total score ranges from 0 to 72 with a higher score indicating greater anxiety sensitivity.
Change in Generalized Anxiety Disorder at weeks 7, 15, and 27 | Week 7, Week 15, Week 27
  Change in Generalized Anxiety Disorder will be assessed with the Generalized Anxiety Disorder 7-item (GAD-7) assessment. GAD-7 total score for the seven items ranges from 0 to 21 where a score ranging from 0-4 indicates minimal anxiety, 5-9 mild anxiety, 10-14 moderate anxiety, and 15-21 severe anxiety.
Change in well-being at weeks 7, 15, and 27 | Week 7, Week 15, Week 27
  Change in well-being will be assessed through the General Life Satisfaction Scale (GLSS). The GLSS total score ranges from 5-35 with higher scores indicating greater life satisfaction.
Anxiety sensitivity as a mediator of treatment effects on PTSD symptoms at week 3 | Week 3
  Anxiety sensitivity will be ascertained with the Anxiety Sensitivity Index-3 (ASI-3). The ASI-3 total score ranges from 0 to 72 with a higher score indicating greater anxiety sensitivity.
App usability at week 3 | Week 3
  App usability which will be ascertained with the System Usability Scale (SUS). The SUS provides a score from 0 to 100. An average SUS score equal to or greater than 68 is considered usable.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States